CLINICAL TRIAL: NCT01381081
Title: A Prospective, Randomized, Double-blinded, Clinical Trial, Comparing Platelet-rich Plasma Intra-articular Knee Injections Versus Corticosteroid Intra-articular Knee Injections for Knee Osteoarthritis
Brief Title: Platelet-rich Plasma Intra-articular Knee Injections for Knee Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRP2010; 2010-023977-21 (EudraCT Number)
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2015-02

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; comparing platelet-rich plasma; intra-articular knee injections
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- platelet-rich plasma intra-articular knee injections (Experimental): a single intra-articular injection of PRP in knee osteoarthritis
  Interventions: Biological: platelet-rich plasma
- Corticosteroid intra-articular knee injections (Active Comparator): a betamethasone and bupivacaine intra-articular injection
  Interventions: Drug: Corticosteroid

INTERVENTIONS:
Biological: platelet-rich plasma — a single intra-articular injection
  Arms: platelet-rich plasma intra-articular knee injections
Drug: Corticosteroid — A single betamethasone and bupivacaine intra-articular injection
  Arms: Corticosteroid intra-articular knee injections

SUMMARY:
The benefit of using platelet rich plasma (PRP) in cartilage injuries, and specifically in degenerative ones, has not been assessed yet. Current studies on the PRP healing or repairing effect on knee cartilage degenerative injuries are not conclusive to establish a standard of behavior, although PRP has shown to improve joint functionality and reduce pain.

Hypothesis: PRP intra-articular injections in osteoarthritic knees reduces pain and leads to a more effective and lasting functional recovering than corticosteroid intra-articular injections.

ELIGIBILITY:
Inclusion Criteria:

* Degenerative osteoarthritis of the knee confirmed radiologically
* Degenerative osteoarthritis of the knee replacement candidate
* Walking ability in patients with or without external support
* Baseline in pain VAS greater than 60

Exclusion Criteria:

* Neoplastic disease
* Immunosuppressive States
* Patients who received intra-articular injections of steroids, anesthetic and / or hyaluronic acid in the last 3 months.
* Patients who have undergone arthroscopic surgery on the last 3 months
* Patients with involvement of bone metabolism except osteoporosis (Paget's disease, renal osteodystrophy, osteomalacia)
* Fibromyalgia or chronic fatigue syndrome
* Liver disease
* Deficit coagulation (blood dyscrasia)
* Thrombocytopenia
* Anticoagulant treatment

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2011-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
The value of the visual analogue scale pain (VAS) | one month after the treatment
  The difference between the baseline and the value of the scale one month after treatment

SECONDARY OUTCOMES:
the value of pain visual analog scale according to | 4 weeks, 3 and 6 months after treatment
the functional level of the knee KOOS | 4 weeks, 3 and 6 months after treatment
All reported adverse events | 4 weeks, 3 and 6 months after treatment
Scale of the SF36 quality of life | 4 weeks, 3 and 6 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nayana Joshi, MD, Principal Investigator — Hospital Vall d'Hebron
Locations (1):
- Hospital Universitario Vall d'Hebron, Barcelona, Barcelona, Spain